CLINICAL TRIAL: NCT03059303
Title: Phase 1, Open-label, Partially Randomized, Parallel-group Study in Healthy Adult Subjects to Assess the Relative Bioavailability of Single-dose Simeprevir (SMV), Odalasvir (ODV), and AL-335 Administered as a Fixed-dose Combination (FDC) Compared With the Single Agents Administered Together, and to Assess the Effect of Multiple-dose Lansoprazole or Omeprazole on the Single-dose Pharmacokinetics of SMV, ODV, and AL-335 Administered as an FDC
Brief Title: Study to Assess the Relative Bioavailability of Fixed-Dose Combination (FDC) Tablet (Simeprevir, Odalasvir and AL-335) Compared With Single Agents Administered Together, and to Assess the Effect of Multiple-Dose Lansoprazole or Omeprazole on Single-Dose Pharmacokinetics of SMV, ODV, and AL-335 (FDC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision to discontinue development of investigational Hep C treatment regimen JNJ-4178: 3 direct acting antivirals - AL-335, ODV & SMV.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108273; 64294178HPC1018 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Healthy
MeSH Terms: interventions — Simeprevir; odalasvir; adafosbuvir; Lansoprazole; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part 1: Treatment A: FDC [SMV(75mg)+ODV(25mg)+AL-335(800mg)] (Experimental): Participants will receive single oral dose of simeprevir (SMV) 75 milligram (mg), odalasvir (ODV) 25 mg, and AL-335 800 mg, given as a fixed-dose combination (FDC) tablet (G008 formulation) after a standardized breakfast on Day 1.
  Interventions: Drug: Simeprevir 75 mg; Drug: Odalasvir 25 mg; Drug: AL-335 800 mg
- Part 1: Treatment B: FDC [SMV(75mg)+ODV(12.5mg)+AL-335(800mg)] (Experimental): Participants will receive single oral dose of SMV 75 mg, ODV 12.5 mg, and AL-335 800 mg, given as an FDC tablet (G007 formulation) after a standardized breakfast on Day 1.
  Interventions: Drug: Simeprevir 75 mg; Drug: Odalasvir 12.5 mg; Drug: AL-335 800 mg
- Part 1: Treatment C: Simeprevir, Odalasvir, and AL-335 (Experimental): Participants will receive single oral dose of 75 mg SMV, 25 mg ODV, and 800 mg AL-335, given as 3 single agents after a standardized breakfast on Day 1.
  Interventions: Drug: Simeprevir 75 mg; Drug: Odalasvir 25 mg; Drug: AL-335 800 mg
- Part 1: Treatment D: Lansoprazole + FDC [SMV+ODV+AL-335] (Experimental): Participants will receive 30 mg lansoprazole once daily in the morning under fasted conditions on Days 1 to 4, and together with a single oral dose of an FDC containing 75 mg SMV, 25 mg ODV, and 800 mg AL-335 (G008 formulation) after a standardized breakfast, which is served 2 hours after lansoprazole dosing, on Day 5.
  Interventions: Drug: Simeprevir 75 mg; Drug: Odalasvir 25 mg; Drug: AL-335 800 mg; Drug: Lansoprazole 30 mg
- Part 1: Treatment E: Omeprazole + FDC [SMV+ODV+AL-335] (Experimental): Participants will receive 20 mg omeprazole once daily in the morning immediately before a (non-standardized) breakfast on Days 1 to 4, and immediately before a standardized breakfast and within 1 hour before a single oral dose of an FDC containing 75 mg SMV, 25 mg ODV, and 800 mg AL-335 (G008 formulation) after a standardized breakfast on Day 5. Treatment E will only be started in case a drug-drug interaction (DDI) is observed for Treatment D.
  Interventions: Drug: Simeprevir 75 mg; Drug: Odalasvir 25 mg; Drug: AL-335 800 mg; Drug: Omeprazole 20 mg
- Part 2: Treatment Sequence A2-F (Experimental): Participants will receive single oral dose of simeprevir (SMV) 75 milligram (mg), odalasvir (ODV) 25 mg, and AL-335 800 mg, given as an FDC (Treatment A2 - G008 formulation) on Day 1 of Period 1, and then single oral dose of SMV 75 mg, ODV 25 mg, and AL-335 800 mg, given as an FDC (Treatment F - G012 formulation) on Day 1 of Period 2, under fed condition (after a standardized breakfast). A washout period of at least 2 weeks will be maintained between each treatment.
  Interventions: Drug: Simeprevir 75 mg; Drug: Odalasvir 25 mg; Drug: AL-335 800 mg
- Part 2: Treatment Sequence F-A2 (Experimental): Participants will receive Treatment F on Day 1 of Period 1 and then Treatment A2 on Day 1 of Period 2 under fed condition (after a standardized breakfast). A washout period of at least 2 weeks will be maintained between each treatment.
  Interventions: Drug: Simeprevir 75 mg; Drug: Odalasvir 25 mg; Drug: AL-335 800 mg
- Part 2: Treatment Sequence C2-F (Experimental): Participants will receive single oral dose of 75 mg SMV, 25 mg ODV, and 800 mg AL-335, given as 3 single agents (Treatment C2) on Day 1 of Period 1 and then Treatment F on Day 1 of Period 2 under fed condition (after a standardized breakfast). A washout period of at least 2 weeks will be maintained between each treatment.
  Interventions: Drug: Simeprevir 75 mg; Drug: Odalasvir 25 mg; Drug: AL-335 800 mg
- Part 2: Treatment Sequence F-C2 (Experimental): Participants will receive Treatment F on Day 1 of Period 1 and then Treatment C2 on Day 1 of Period 2 under fed condition (after a standardized breakfast). A washout period of at least 2 weeks will be maintained between each treatment.
  Interventions: Drug: Simeprevir 75 mg; Drug: Odalasvir 25 mg; Drug: AL-335 800 mg
- Part 2: Treatment Sequence C2-G (Experimental): Participants will receive Treatment C2 on Day 1 of Period 1 and then 2 tablets of SMV 37.5 mg, ODV 37.5 mg, and AL-335 400 mg, given as FDC (Treatment G - G013 formulation) on Day 1 of Period 2 under fed condition (after a standardized breakfast). A washout period of at least 2 weeks will be maintained between each treatment.
  Interventions: Drug: Simeprevir 75 mg; Drug: Odalasvir 25 mg; Drug: Odalasvir 75 mg; Drug: AL-335 800 mg
- Part 2: Treatment Sequence G-C2 (Experimental): Participants will receive Treatment G on Day 1 of Period 1 and then Treatment C2 on Day 1 of Period 2 under fed condition (after a standardized breakfast). A washout period of at least 2 weeks will be maintained between each treatment.
  Interventions: Drug: Simeprevir 75 mg; Drug: Odalasvir 25 mg; Drug: Odalasvir 75 mg; Drug: AL-335 800 mg
- Part 2: Treatment Sequence F-G (Experimental): Participants will receive Treatment F on Day 1 of Period 1 and then Treatment G on Day 1 of Period 2 under fed condition (after a standardized breakfast). A washout period of at least 2 weeks will be maintained between each treatment.
  Interventions: Drug: Simeprevir 75 mg; Drug: Odalasvir 25 mg; Drug: Odalasvir 75 mg; Drug: AL-335 800 mg
- Part 2: Treatment Sequence G-F (Experimental): Participants will receive Treatment G on Day 1 of Period 1 and then Treatment F on Day 1 of Period 2 under fed condition (after a standardized breakfast). A washout period of at least 2 weeks will be maintained between each treatment.
  Interventions: Drug: Simeprevir 75 mg; Drug: Odalasvir 25 mg; Drug: Odalasvir 75 mg; Drug: AL-335 800 mg

INTERVENTIONS:
Drug: Simeprevir 75 mg — Part 1: Simeprevir (SMV) 75 mg taken orally as a component of FDC tablet in Treatment A, B, D and E and as a single agent capsule in Treatment C.
  Part 2: SMV 75 mg taken orally as a component of FDC tablet in Treatment A2, F (2 tablets of 37.5 mg each), and G (2 tablets of 37.5 mg each), and as a single agent capsule in Treatment C2.
Drug: Odalasvir 25 mg — Part 1: Odalasvir (ODV) 25 mg taken orally as a component of FDC tablet in Treatment A, D and E and as a single agent tablet in Treatment C.
  Part 2: ODV 25 mg taken orally as a component of FDC tablet in Treatment A2 and F (2-tablets of 12.5 mg each), and as a single agent tablet in Treatment C2.
  Arms: Part 1: Treatment A: FDC [SMV(75mg)+ODV(25mg)+AL-335(800mg)]; Part 1: Treatment C: Simeprevir, Odalasvir, and AL-335; Part 1: Treatment D: Lansoprazole + FDC [SMV+ODV+AL-335]; Part 1: Treatment E: Omeprazole + FDC [SMV+ODV+AL-335]; Part 2: Treatment Sequence A2-F; Part 2: Treatment Sequence C2-F; Part 2: Treatment Sequence C2-G; Part 2: Treatment Sequence F-A2; Part 2: Treatment Sequence F-C2; Part 2: Treatment Sequence F-G; Part 2: Treatment Sequence G-C2; Part 2: Treatment Sequence G-F
Drug: Odalasvir 12.5 mg — Part 1: ODV 12.5 mg taken orally as a component of FDC tablet in Treatment B.
  Arms: Part 1: Treatment B: FDC [SMV(75mg)+ODV(12.5mg)+AL-335(800mg)]
Drug: Odalasvir 75 mg — Part 2: ODV 75 mg taken orally as a component of FDC tablet (2 tablets of 37.5 mg each) in Treatment G.
  Arms: Part 2: Treatment Sequence C2-G; Part 2: Treatment Sequence F-G; Part 2: Treatment Sequence G-C2; Part 2: Treatment Sequence G-F
Drug: AL-335 800 mg — Part 1: AL-335 800 mg taken orally as a component of FDC tablet in Treatment A, B, D and E and as a single agent tablet in Treatment C.
  Part 2: AL-335 800 mg taken orally as a component of FDC tablet in Treatment A2, F (2 tablets of 400 mg each), and G (2 tablets of 400 mg each) and as a single agent tablet in Treatment C2.
Drug: Lansoprazole 30 mg — 30 mg lansoprazole once daily from Day 1 to Day 5.
  Other Names: Prevacid
  Arms: Part 1: Treatment D: Lansoprazole + FDC [SMV+ODV+AL-335]
Drug: Omeprazole 20 mg — 20 mg omeprazole once daily from Day 1 to Day 5.
  Arms: Part 1: Treatment E: Omeprazole + FDC [SMV+ODV+AL-335]

SUMMARY:
The purpose of this study is to assess the relative bioavailability of single-dose Simeprevir (SMV), Odalasvir (ODV), and AL-335 when administered as a fixed-dose combination (FDC) compared with the single agents when administered together, and to assess the effect of multiple-dose lansoprazole and omeprazole on the single-dose pharmacokinetics (PK) of SMV, ODV, and AL-335 when administered as an FDC.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a body mass index (BMI: weight in kg divided by the square of height in meters) of 18.0 to 32.0 kilogram per meter (kg/m^2), extremes included, and a body weight not less than 50.0 kg
* Participant must have a blood pressure (supine after at least 5 minutes rest) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic. If blood pressure is out of range, up to 2 repeated assessments are permitted. Participants with a normal value at retest may be included
* Participant must have a normal 12-lead Electrocardiogram [ECG] (based on the mean value of triplicate ECG parameters) consistent with normal cardiac conduction and function at screening, including:a) normal sinus rhythm (heart rate (HR) between 60 and 90 beats per minute [bpm], extremes included); b) QT interval corrected for heart rate according to Fridericia's formula (QTcF) less than or equal to <=450 milliseconds (ms) for male participants and <=470 ms for female participants; c) QRS interval <=110 ms; d) PR interval <=200 ms; e) Electrocardiogram (ECG) morphology consistent with healthy cardiac conduction and function. Any evidence of heart block is exclusionary. Any evidence of left or right bundle branch block is exclusionary
* Female participant must have a negative highly sensitive urine or serum pregnancy test at Day -1

Exclusion Criteria:

* Participant with a past history of: a) Heart arrhythmias (example, extrasystolic rhythms or tachycardia at rest). Isolated extrasystolic beats are not exclusionary; b) Risk factors associated with Torsade de Pointes such as hypokalemia; c) Family history of short/long QT syndrome; d) Sudden unexplained death (including sudden infant death syndrome) in a first degree relative (that is, sibling, offspring, or biological parent)
* Participant has known allergies, hypersensitivity, or intolerance to odalasvir (ODV), AL-335, simeprevir (SMV), lansoprazole, or omeprazole, or their excipients
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at screening
* Participant has a history of human immunodeficiency virus (HIV-1) or -2 infection positive, or tests positive for HIV-1 or -2 at screening
* Participant has previously been dosed with SMV, ODV, or AL-335 in more than 3 single-dose studies or in a multiple dose study with SMV, ODV, or AL-335

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

PRIMARY OUTCOMES:
Part 1: Maximum Observed Plasma Concentration (Cmax) of Simeprevir (SMV) | Predose, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 hours post-dose
  Cmax is defined as the maximum observed plasma concentration.
Part 2: Maximum Observed Plasma Concentration (Cmax) of SMV | Predose, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 hours post-dose
  Cmax is defined as the maximum observed plasma concentration.
Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Quantifiable (AUC [0-last]) of SMV | Predose, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 hours post-dose
  AUC (0-last) is the area under the plasma concentration-time curve (AUC) from time 0 to the time of the last measurable (non below quantification limit [non BQL]) concentration, calculated by linear trapezoidal summation.
Part 2: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Quantifiable (AUC [0-last]) of SMV | Predose, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 hours post-dose
  AUC (0-last) is the area under the plasma concentration-time curve (AUC) from time 0 to the time of the last measurable (non below quantification limit [non BQL]) concentration, calculated by linear trapezoidal summation.
Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of SMV | Predose, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 hours post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time calculated as the sum of AUC (0-last) and C (0-last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(0-last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant.
Part 2: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of SMV | Predose, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 hours post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time calculated as the sum of AUC (0-last) and C (0-last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(0-last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant.
Part 1: Maximum Observed Plasma Concentration (Cmax) of Odalasvir (ODV) | Predose, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 288, 312 hours post-dose
  Cmax is defined as the maximum observed plasma concentration.
Part 2: Maximum Observed Plasma Concentration (Cmax) of ODV | Predose, 1, 2, 4, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 288, and 312 hours post-dose
  Cmax is defined as the maximum observed plasma concentration.
Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Quantifiable (AUC [0-last]) of ODV | Predose, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 288, 312 hours post-dose
  AUC (0-last) is the area under the plasma concentration-time curve (AUC) from time 0 to the time of the last measurable (non below quantification limit [non BQL]) concentration, calculated by linear trapezoidal summation.
Part 2: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Quantifiable (AUC [0-last]) of ODV | Predose, 1, 2, 4, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 288, and 312 hours post-dose
  AUC (0-last) is the area under the plasma concentration-time curve (AUC) from time 0 to the time of the last measurable (non below quantification limit [non BQL]) concentration, calculated by linear trapezoidal summation.
Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of ODV | Predose, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 288, 312 hours post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time calculated as the sum of AUC (0-last) and C (0-last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration time curve from time zero to last quantifiable time, C(0-last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant.
Part 2: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of ODV | Predose, 1, 2, 4, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 288, and 312 hours post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time calculated as the sum of AUC (0-last) and C (0-last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration time curve from time zero to last quantifiable time, C(0-last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant.
Part 1: Maximum Observed Plasma Concentration (Cmax) of AL-335 | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  Cmax is defined as the maximum observed plasma concentration.
Part 2: Maximum Observed Plasma Concentration (Cmax) of AL-335 | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  Cmax is defined as the maximum observed plasma concentration.
Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Quantifiable (AUC [0-last]) of AL-335 | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  AUC (0-last) is the area under the plasma concentration-time curve (AUC) from time 0 to the time of the last measurable (non below quantification limit [non BQL]) concentration, calculated by linear trapezoidal summation.
Part 2: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Quantifiable (AUC [0-last]) of AL-335 | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  AUC (0-last) is the area under the plasma concentration-time curve (AUC) from time 0 to the time of the last measurable (non below quantification limit [non BQL]) concentration, calculated by linear trapezoidal summation.
Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of AL-335 | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time calculated as the sum of AUC (0-last) and C (0-last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration time curve from time zero to last quantifiable time, C(0-last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant.
Part 2: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of AL-335 | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time calculated as the sum of AUC (0-last) and C (0-last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration time curve from time zero to last quantifiable time, C(0-last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant.
Part 1: Analyte Concentration at 1 Hour Post Dosing (C1h) of Lansoprazole | Day 5 (1 hour post dose)
  Analyte Concentration at 1 Hour Post Dosing (C1h) of Lansoprazole
Part 1: Analyte Concentration at 2 Hour Post Dosing (C2h) of Lansoprazole | Day 5 (2 hour post dose)
  Analyte Concentration at 2 Hour Post Dosing (C2h) of Lansoprazole.
Part 1: Analyte Concentration at 1 Hour Post Dosing (C1h) of Omeprazole (if applicable) | Day 5 (1 hour post dose)
  Analyte concentration will only be assessed if participants receive omeprazole (only in case a drug-drug interaction [DDI] is observed for participants who received lansoprazole).
Part 1: Analyte Concentration at 2 Hour Post Dosing (C2h) of Omeprazole (if applicable) | Day 5 (2 hour post dose)
  Analyte concentration will only be assessed if participants receive omeprazole (only in case an DDI is observed for participants who received lansoprazole).

SECONDARY OUTCOMES:
Part 2: Exposure as Measured by AUC From 2 Different Fixed Dose Combination Formulations containing odalasvir (ODV) (Treatment F Versus Treatment A2) | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  Exposure will be measured by AUC.
Part 1 and 2: Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Screening (21 days prior to the first dose) to follow up Phase (30 to 35 days after last dose)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, irrespective of a causal relationship with the investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Celerion, Tempe, Arizona, United States